CLINICAL TRIAL: NCT05944484
Title: Effect of Visceral vs Total Body Fat Reduction in Obese Female With Stress Urinary Incontinence by EMG and Iciq Questionnaire
Brief Title: Effect of Visceral vs Total Body Fat Reduction in Obese Female With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dina Mohamed Tarek Mansour El-kasrawy (Other)
Responsible Party: Sponsor-Investigator, Dina Mohamed Tarek Mansour El-kasrawy, physiotherapist at EL-AHRAR teaching hospital, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Effect of fat on SUI
Record Dates: First submitted 2023-06-11; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Stress Urinary Incontinence
Keywords: Visceral fat; total body fat; obese female; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Visceral fat reduction vs total body fat reduction on obese female with stress urinary incontinence
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (participant,outcomes Assessor) Random generator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- kegel exercises (Active Comparator): Kegel exercise program performed for 12 weeks( 3 sessions /week )
  .• "The first step is external observation, with the patient in the lithotomy position.And describe for each woman how to feel her muscle when she stops mid-stream urine.
  * "The second step is vaginal examination, performed gently with one finger." - The digital exam served a double purpose: first to assess the development of the puboccocygeus muscle and second to verify that the patient was able to identify the correct muscle
  * The third stage main exercises quick flick : contract muscle as quickly as possible 10-20 times then relax then count 10 for relax then reapeat .( 50 repetitions) slow contraction: tighten the muscle as hard as you can for account of 10 -20 .relax for acount 10 then repeat ( 50 repetitions) sustained contraction: tighten the muscle halfway and hold 60 seconds .relax for account 20 then repeat (10 repetitions)
  Interventions: Behavioral: low caloric diet, ultrasound cavitation,Kegel exercises
- low caloric diet (Active Comparator): low caloric diet (800-1200) calories/day . According to each patient, diet should contain (carbohydrate protein, fats, minerals, vitamins),1200 calories in the first month, 1000 calories in the second month, and 800 calories in the third month. Every week, each woman will be allowed to change the types of food to avoid boarding.
  Interventions: Behavioral: low caloric diet, ultrasound cavitation,Kegel exercises
- ultrasound cavitation (Active Comparator): ultrasound cavitation, for 30 minutes on abdomen with continuous emission and frequency of 40 KHz, 3-6 W/cm2, 60W with 10cm2 active surface, twice/ week with 3 days apart for 12 weeks.
  Interventions: Behavioral: low caloric diet, ultrasound cavitation,Kegel exercises

INTERVENTIONS:
Behavioral: low caloric diet, ultrasound cavitation,Kegel exercises — * low caloric diet (800-1200) calories/day,). According to each patient, diet contained (carbohydrate protein, fats, minerals, vitamins). 50 to 55% of total calories are carbohydrates, 10 to 15% of total calories protein. Fat limited to less than about 28% of daily total calories .Women took 1200 calories in the first month, 1000 calories in the second month, and 800 calories in the third month. Every week, each woman allowed to change the types of food to avoid boarding.
  * ultrasound cavitation emits low-frequency ultrasound 40 khz for 30 minutes on abdomen twice/ week with 3 days apart for 12 weeks.
  kegel exercise: Each woman in the study took the same Kegel exercise program performed the Kegel exercise for 12 weeks (3 sessions per week)

SUMMARY:
The aim of this study is to investigate the visceral fat reduction versus total body fat reduction on stress urinary incontinence in obese females.

DETAILED DESCRIPTION:
compare the effect of visceral fat reduction versus total body fat reduction on stress urinary incontinence in obese females.

control group: consist of 20 obese women. They will receive Kegel exercises only 3 session/ week for 12 weeks.

Diet group: consist of 20 obese women. They will receive low caloric diet and Kegel exercises 3 session/week for 12 weeks.

Ultrasound cavitation group: consist of 20 obese women. They will receive Kegel exercises 3 session/week and ultrasound cavitation two sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* They will be diagnosed with stress urinary incontinence grade≥ 1
* Their age will range from 35-48 years old.
* Their body mass index will exceed 29.9 kg/m².
* Their hip waist ratio will be more than 0.85 cm.
* They will be multipara >1.

Exclusion Criteria:

* · Fecal incontinence, urge incontinence, overflow incontinence or functional incontinence or prolapse.

  * Diabetes, asthma, cardiovascular, or renal diseases
  * Taking medication for stress urinary incontinence or hormonal replacement therapy.
  * Gynecological surgeries, or surgeries for obesity.
  * Pregnant women.

Ages: 35 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Obese female
Enrollment: 60 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
stress urinary incontinence | 12 weeks
  evaluate stress urinary incontinence by The International Consultation on Incontinence Questionnaire ranged from (0-21)
  Question items:
  Frequency or urinary incontinence Amount of leakage Overall impact of urinary incontinence Self-diagnostic item. The ICIQ-UI Short form provides a score ranging from 0-21. With a higher score indicating greater severity of symptoms. The "self-diagnostic" portion of the questionnaire is not given a score

SECONDARY OUTCOMES:
waist circumference | 12 weeks
  measure waist circumference in centimeter
Measure weight | 12 weeks
  Measure weight in kilogram
Measure body mass index | 12 weeks
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No